CLINICAL TRIAL: NCT06994065
Title: Efficacy of Ferric Carboxymaltose Versus Iron Sucrose in Non-dialysis Dependent Chronic Kidney Disease Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sindh Institute of Urology and Transplantation (Other)
Responsible Party: Principal Investigator, Kamlesh Kumar, FCPS Nephrology Resident, Sindh Institute of Urology and Transplantation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRONEASE Trial
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Iron Deficiency Anemia Associated With Non-Dialysis Dependent Chronic Kidney Disease
MeSH Terms: interventions — ferric carboxymaltose; Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ferric Carboxymltose (FCM) (Experimental): Participants will receive intravenous Ferric Carboxymaltose according to their Iron deficit
  Interventions: Drug: Ferric Carboxymaltose (FCM)
- Iron Sucrose (IS) (Experimental): Participants will receive intravenous Iron Sucrose according to their Iron deficit
  Interventions: Drug: Iron Sucrose injection

INTERVENTIONS:
Drug: Ferric Carboxymaltose (FCM) — This study will dose each patient according to their calculated iron deficit through Ganozi formula Iron deficit(mg) = bodyweight(kg) x (target Hb - actual Hb) (g/dl) x 2.4 + Iron storage depot(mg)
  Other Names: Ferric Carboxy maltose; Ferinject
  Arms: Ferric Carboxymltose (FCM)
Drug: Iron Sucrose injection — This study will dose each patient according to their calculated iron deficit through Ganozi formula Iron deficit(mg) = bodyweight(kg) x (target Hb - actual Hb) (g/dl) x 2.4 + Iron storage depot(mg)
  Other Names: Venofer
  Arms: Iron Sucrose (IS)

SUMMARY:
The goal of this clinical trial is to learn if Ferric Carboxymaltose is a safe efficacious alternative to Iron Sucrose for treatment of Iron deficiency anemia in non-dialysis dependent chronic kidney disease patients. The main questions it aims to answer are:

* Does Ferric Carboxymaltose causes similar or higher rise in hemoglobin concentration and serum Ferritin and transferrin saturation
* What medical problems will participants have when receiving Ferric Carboxymaltose

Participants will:

* Be administered either Ferric Carboxymaltose or Iron Sucrose
* Visit the clinic at day 28 and 56 for checkup and tests
* Be monitored for any medical problem during and after infusion

DETAILED DESCRIPTION:
Anemia is a common complication of chronic kidney disease with its prevalence increasing with disease progression. The major causes of anemia in patients who have CKD are iron and erythropoietin deficiency. For management of iron deficiency either oral or intravenous iron products are used. Currently Iron Sucrose is being used as drug of choice for intravenous iron replacement for treatment of iron deficiency anemia as standard of care in Pakistan.

Objective of this study is to compare Ferric Carboxymaltose versus Iron Sucrose for treatment of iron deficiency anemia.

This study will be conducted at the department of Nephrology, Sindh Institute of Urology and Transplantation (SIUT), Karachi, Sindh, Pakistan. Data will be collected after taking approval of Institutional review board and Ethical review Committee and informed written consent from the participants.

Participants will be enrolled by principal investigator. All participants will be randomized into two groups by sealed envelopes.

After enrollment, participants will be administered either Ferric Carboxymaltose or Iron Sucrose at daycare clinic of department, Dose will be according to calculated iron deficit though Ganozi formula. Iron deficit(mg) = bodyweight(kg) x (target hemoglobin - actual hemoglobin ) (g/dl) x 2.4 + Iron storage depot(mg).

Medical problems (adverse effects) will be monitored, noted and treated accordingly.

Laboratory parameters such as hemoglobin, serum ferritin and transferrin saturation will be checked at baseline and scheduled visits, which will be compared at the end of study.

After completion of data collection, data analysis will be done using Statistical package for social sciences 26.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Between age 18-85 years
* Patients diagnosed with Chronic kidney disease having eGFR of less than 60 ml/kg/1.73m2 (not on maintenance dialysis)

Exclusion Criteria:

* Patients on maintenance dialysis
* Patients with concomitant B12 or folate deficiency
* Patients receiving ESA therapy
* Patients with prior Iron replacement therapy within preceding 2 weeks
* Patients receiving blood transfusions within preceding 3 months
* Pregnant Females
* Patients with Upper GI Bleeding
* Patients with history of hematologic disorders, active malignancy or chronic inflammatory conditions like tuberculosis or ulcerative colitis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in hemoglobin concentration | Baseline, Day 28, Day 56
Change from baseline in Transferrin Saturation (TSAT) | Baseline, Day 28, Day 56
  Transferrin Saturation (TSAT) will be calculated as:
  TSAT (%) = 100 x Serum Iron/Total Iron binding capacity (TIBC)
Change from baseline in serum Ferritin | Baseline, Day 28, Day 56

SECONDARY OUTCOMES:
Safety, as measured by number of subjects with at least one adverse event | Baseline, Day 28, Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Kamlesh Kumar, MBBS, (FCPS Resident), Principal Investigator — Sindh Institute of Urology and Transplantaion
Locations (1):
- Sindh Institute of Urology and Transplantaion, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Szczech LA, Bregman DB, Harrington RA, Morris D, Butcher A, Koch TA, Goodnough LT, Wolf M, Onken JE. Randomized evaluation of efficacy and safety of ferric carboxymaltose in patients with iron deficiency anaemia and impaired renal function (REPAIR-IDA): rationale and study design. Nephrol Dial Transplant. 2010 Jul;25(7):2368-75. doi: 10.1093/ndt/gfq218. Epub 2010 Apr 21. PMID 20466657
- [Result] Onken JE, Bregman DB, Harrington RA, Morris D, Buerkert J, Hamerski D, Iftikhar H, Mangoo-Karim R, Martin ER, Martinez CO, Newman GE, Qunibi WY, Ross DL, Singh B, Smith MT, Butcher A, Koch TA, Goodnough LT. Ferric carboxymaltose in patients with iron-deficiency anemia and impaired renal function: the REPAIR-IDA trial. Nephrol Dial Transplant. 2014 Apr;29(4):833-42. doi: 10.1093/ndt/gft251. Epub 2013 Aug 20. PMID 23963731
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/23963731/